CLINICAL TRIAL: NCT03742817
Title: Effects of e-Cigarettes on Perceptions and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Professor of Preventive Medicine, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HS-18-00839 - Pilot Study
Record Dates: First submitted 2018-11-14; First posted 2018-11-15 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Electronic Cigarettes
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sweet-Flavor 4.5% Nicotine (Salt) (Experimental): Participants will self-administer a sweet-flavored e-cigarette containing 4.5% nicotine by volume.
  Interventions: Other: e-Cigarette
- Sweet-Flavor 0 mg/mL Nicotine (Free-Base) (Placebo Comparator): Participants will self-administer a sweet-flavored e-cigarette containing 0 mg/mL nicotine.
  Interventions: Other: e-Cigarette
- Sweet-Flavor 6 mg/mL Nicotine (Free-Base) (Experimental): Participants will self-administer a sweet-flavored e-cigarette containing 6 mg/mL nicotine.
  Interventions: Other: e-Cigarette
- Usual e-Cigarette (Active Comparator): Participants will self-administer either their preferred brand combustible cigarette or e-cigarette with usual nicotine nicotine concentration.
  Interventions: Other: e-Cigarette

INTERVENTIONS:
Other: e-Cigarette — Participants will self-administer an experimenter-provided e-cigarette.

SUMMARY:
This project will assess the ways in which e-cigarette product diversity impacts the user experience to inform potential regulations by identifying product characteristics that may: (1) put young adults at risk for tobacco product use; and (2) facilitate adult smokers switching to e-cigarettes. There are three primary objectives to the study: (1) Determine which dimensions of e-cigarette product diversity differentially affect product appeal across young adult e-cigarette users and middle-age/older adult smokers with an interest in, but no significant experience with, e-cigarettes; (2) Determine which dimensions of e-cigarette product diversity differentially affect abuse liability in young adult e-cigarette users and the ability to resist smoking in adult smokers with an interest in, but no significant experience with, e-cigarettes; (3) Determine the affect of product characteristics on e-cigarette nicotine delivery profile. For Aim 1, young adult vapers (N=200) and adult smokers (N=200) will attend one laboratory session in which they will self-administer e-cigarette products varied according to within-subject e-cigarette factors (e.g., flavor, pg/vg ratio). For Aim 2, young adults vapers (N=360) and adult smokers (N=360) will administer an e-cigarette product and complete behavioral economic tasks that test the participant's choice of earning money to delay initiation and continued use of: (1) The sampled e-cigarette product (abuse liability; young adult vapers); or (2) Their own brand cigarettes (ability to resist smoking; adult current smokers). A pilot study will establish device and e-liquid parameters (e.g., nicotine concentration) to be used for all aims.

ELIGIBILITY:
Inclusion Criteria:

Vapers

1. E-cigarette use >3 day/week for >2 months
2. Report regularly using e-cigarette products with nicotine
3. Positive cotinine test via NicAlert test strip

Smokers

1. Daily cigarette smoking for ≥ 2 years
2. Currently smoke > 4 cig/day
3. Interest in trying an e-cigarette or current use of e-cigarettes

Exclusion Criteria:

Vapers

1. Pregnancy/breastfeeding
2. Desire to immediately reduce e-cigarette use

Smokers

1. Breath CO < 9ppm at intake
2. Pregnancy / breastfeeding
3. Current daily use of other combustible tobacco products (e.g., cigars)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Subjective Appeal | 1 hour
  Self-report measures of product appeal will be completed following the e-cigarette administration.
Positive Affect Negative Affect Schedule | 4 hours
  The 10-item Positive Affect Negative Affect Schedule (PANAS-SF) will be used to measure positive and negative affect.
Questionnaire of Vaping Urges | 4 hours
  10-item Brief Questionnaire of Vaping Urges will assess desire, intention, urge and need to vape e-cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Leventhal, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han DH, Wong M, Peraza N, Vogel EA, Cahn R, Mason TB, Kirkpatrick M, Tackett AP, Leventhal AM. Dose-response effects of two nicotine salt formulations on electronic cigarette appeal and sensory attributes. Tob Control. 2023 Jan 2:tobaccocontrol-2022-057553. doi: 10.1136/tc-2022-057553. Online ahead of print. PMID 36593119